CLINICAL TRIAL: NCT03797053
Title: Expansion ex Vivo Des Cellules Tumorales Circulantes Comme modèle de Pharmacologie prédictive Des Cancers. EXPEVIVO-CTC
Brief Title: Ex Vivo Expansion of Circulating Tumor Cells as a Model for Cancer Predictive Pharmacology
Acronym: EXPEVIVO-CTC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ScreenCell (Industry); Celenys (Unknown); Imstar (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI15009
Record Dates: First submitted 2018-03-09; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-03

CONDITIONS: Melanoma; Circulating Tumor Cell
MeSH Terms: conditions — Melanoma; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood Sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 : metastatic cohort: Cohort1: Cohort of patients with stage III inoperable or IV metastatic melanoma This cohort will enable the achievement of objectives 1 (proof of concept) and 2 (establishment of prognostic and predictive value).
  Interventions: Procedure: Biological sample
- Cohort 2 : adjuvant cohort: Cohort 2: Cohort of patients with melanoma who are candidates for sentinel lymph node analysis.
  This group includes patients with melanoma in whom sentinel lymph node testing is performed. According to current French recommendations, these are patients whose primary melanoma has a Breslow index (thickness) of more than 1 mm or ulcerated primary melanoma (loss of the epidermis).
  Interventions: Procedure: Biological sample

INTERVENTIONS:
Procedure: Biological sample — Biological sample performed :
  * before treatment
  * 1 months after the beginning of treatment
  * every tumoral assessment

SUMMARY:
Several studies conducted over the past decade have shown that Circulating tumor cells (CTCs) can be used as a marker for predicting disease progression and survival in patients with early or metastatic cancer. A high number of CTCs correlate with aggressive disease, increased metastasis and decreased survival rates.

Knowledge of metastasis mechanisms was mainly obtained from mouse models with CTCs after orthotopic transplants. The only possibility to study the patient's CTC subpopulations is to carry out ex-vivo expansion and develop an animal model with CTC xenograft. Because circulating blood collection is simple and non-invasive, CTCs can be used as a marker to track disease progression and survival in real time. CTCs could also guide therapeutic choice.

ELIGIBILITY:
COHORT 1

Inclusion Criteria:

* Histologically confirmed cutaneous or mucosal melanoma (per American joint committee on cancer (AJCC) staging system) that is unresectable or metastatic
* No prior systemic anticancer therapy for unresectable/metastatic melanoma or clinical/radiological disease progression (RECIST1.1) if previously treated and before new treatment
* No prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as cutaneous carcinoma or cervix)
* followed in Saint Louis Hospital
* Tumor tissue available in Saint Louis Hospital
* Subjects must have signed and approved written informed consent form
* No pregnancy
* Any positive test for hepatitis A virus, hepatitis B virus or hepatitis C virus indicating acute or chronic infection, and/or detectable virus

Exclusion Criteria:

* None

COHORT 2 :

Inclusion Criteria :

* Histologically confirmed cutaneous or mucosal melanoma
* Candidates for sentinel lymph node analysis and surgical recovery (this examination is in practice reserved for melanomas >1mm thick or ulcerated)
* No prior adjuvant anticancer therapy
* followed in Saint Louis Hospital
* Tumor tissue available in Saint Louis Hospital
* Subjects must have signed and approved written informed consent form
* No pregnancy
* Any positive test for hepatitis A virus, hepatitis B virus or hepatitis C virus indicating acute or chronic infection, and/or detectable virus

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort1: Cohort of patients with stage III unresectable or IV metastatic melanoma patients Cohort 2: Cohort of patients with melanoma candidates for sentinel lymph node analysis
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2015-04-06 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Therapeutical response | 6 months
  Occurrence of clinical benefit (defined as Complete Response (CR), Partial Response (PR) or stable disease (SD)) and progressive disease based on the best overall response which depends on the tumour evaluations assessed using RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Survival | 1 year
Survival | 3 years
Survival | 5 years
Disease free Survival | 1 year
Disease free Survival | 3 years
Disease free Survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No